CLINICAL TRIAL: NCT01465165
Title: Comparison of Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) and Magnetic Resonance Spectroscopy (MRS) as Bioenergetic Imaging Modalities in Healthy Human Brain and Major Depressive Disorder
Brief Title: Use of Multiple Brain Imaging Modalities (PET and MRS) to Identify Metabolic Abnormalities in Major Depression
Status: Terminated | Type: Observational
Why Stopped: Study procedures were not feasible.
Sponsor: Paul Carlson (Other)
Collaborators: Western Institute for Biomedical Research (Unknown); University of Utah (Other); Molecular Imaging Program, Huntsman Cancer Institute (Unknown)
Responsible Party: Sponsor-Investigator, Paul Carlson, Assistant Professor, University of Utah
Organization: University of Utah (Other)
Other Study IDs: WIBR08-PJC
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Positron emission tomography; Magnetic resonance spectroscopy; glucose metabolism; ATP; phosphocreatine
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Depressed, unmedicated: Participants with MDD who are not treated with any antidepressant medication
- Depressed, on antidepressant: Participants with MDD, currently depressed but on a stable dose of an SSRI antidepressant
- Healthy control: Healthy participant with no MDD or other psychiatric condition, matched by age and gender to MDD participants

SUMMARY:
Several lines of evidence support the existence of an underlying abnormality in brain energy metabolism may play a key role in the biology of mood disorders. The current study utilizes two distinct but complementary imaging techniques, fluorodeoxyglucose (FDG) positron emission tomography (PET) and multinuclear magnetic resonance spectroscopy (MRS), to better understand the nature of these metabolic abnormalities in major depressive disorder (MDD). The investigators hypothesize that individuals with depression will have increased metabolic activity as measured by PET in certain brain regions involved in mood regulation, but that this metabolic activity will be inefficient based on MRS findings. For this study, the investigators will study 10 medication-free, currently depressed participants with recurrent MDD, 10 depressed participants with recurrent MDD currently taking antidepressant medication, and up to 20 healthy control participants matched to depressed participants for age and gender. Depressed and healthy participants will each undergo one PET scan and one MRS scanning session.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for Major Depressive Disorder (MDD), Recurrent
* Montgomery-Asberg Depression Rating Scale (MADRS) score > 18

Exclusion Criteria:

* Any coexisting psychiatric illness other than generalized anxiety disorder, panic disorder, or social/specific phobias
* Any history of substance dependence
* Substance abuse within the past 6 months
* Significant risk of suicide, as defined by score >4 on item 10 of the MADRS or in the clinical judgment of the study physician
* Any significant medical or neurological condition which is likely to impact the central nervous system and/or affect the results of MRS or PET imaging
* For the subset of unmedicated MDD patients, any psychotropic medications within 4 weeks prior to scanning. For the subgroup of medicated patients, they may be taking a stable dose (i.e., same dose for at least 4 weeks at the time of scanning) of standard antidepressant medications, but may not be taking any other psychotropic medication.
* Inability to give informed consent
* Contraindication to MRI (e.g., pacemaker, ferromagnetic implants in the body)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-05-15 (Actual); Primary Completion 2012-06-24 (Actual); Study Completion 2012-06-24 (Actual)

PRIMARY OUTCOMES:
high energy phosphate metabolites (Phosphocreatine (PCr)) as measured by magnetic resonance spectroscopy | cross-sectional
  relative concentration of Pcr

SECONDARY OUTCOMES:
regional cerebral glucose metabolism, as measured by Positron Emission Tomography (PET) | cross-sectional
  binding potential of FDG
N-Acetyl-Aspartate (NAA) metabolite intensity, as measured by proton Magnetic Resonance Spectroscopy (MRS) | cross-sectional
  relative concentration of NAA
severity of depressive symptoms, as scored on the Montgomery-Asberg Depression Rating Scale (MADRS) | cross-sectional
  MADRS composite score

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Carlson, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Dept of Psychiatry, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified scanning images may be individually examined after the study is completed if new analysis methods become available to collaborators.